CLINICAL TRIAL: NCT07166302
Title: Ultrasound Evaluation of Hematoma Risk After Needle EMG in Patient on DOAC Therapy
Acronym: U-HAND
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: University Hospital Brno (Unknown)
Responsible Party: Principal Investigator, Adam Betik, MD, Masaryk University
Other Study IDs: 870177; PIG I/22 (Other Grant/Funding Number: University Hospital Brno)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Direct Acting Anticoagulant Adverse Reaction; Needle Injury; EMG; Peripheral Neuropathies; Mononeuropathies; Polyneuropathies; Neuromuscular Diseases (NMD)
Keywords: electromyography; hematoma; ultrasonography; anticoagulants
MeSH Terms: conditions — Peripheral Nervous System Diseases; Mononeuropathies; Polyneuropathies; Neuromuscular Diseases; Hematoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOAC patients: Patients using direct anticoagulants and undergoing needle EMG for whatever reason

SUMMARY:
Approximately 30 minutes after needle EMG, patients who are taking direct oral anticoagulants (DOACs) will undergo an ultrasound examination to evaluate for the presence of possible intramuscular hematomas at the muscles where the EMG needle was inserted. These hematomas are considered a potential adverse effect of needle EMG.

The aim of the study is to determine whether needle EMG can be considered a safe procedure in this group of patients, without posing a risk of intramuscular hematoma formation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must understand the nature of the study and must provide signed and dated written informed consent prior to conducting any study-related procedures
* Willing and able to comply with all protocol procedures
* subjects confirmed the daily (and recent) intake od direct anticoagulants in strandard dosing.
* no other antitrombotic drug therapy (e.g. acetylsalicyl acid, clopidogrel, ticagralol, low molecular weight heparin or second direct anticoagulant) is taken.

Exclusion Criteria:

* Any clinically significant medical or psychiatric condition or medical history that, in the opinion of the investigator, would interfere with the subject's ability to participate in the study or increase the risk of participation for that subject
* other antitrombotic drug therapy (e.g. acetylsalicyl acid, clopidogrel, ticagralol, low molecular weight heparin or second direct anticoagulant) is recently taken.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing needle EMG examination in EMG laboratory
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intramuscular hematoma risk | seven days since the needle EMG
  Ultrasound evaluation of intramuscular hematoma formation after needle EMG in DOAC patients

CONTACTS AND LOCATIONS:
Overall Officials: Eva Vlckova, MD, Study Chair — Masaryk University, University Hospital Brno
Locations (2):
- Czechia (2):
  - University Hospital Brno, Brno, Czech Republic
  - University hospital Brno, Brno, Czech Republic

IPD SHARING:
Plan to Share IPD: No